CLINICAL TRIAL: NCT04281992
Title: A Phase 1/2A Clinical Study to Evaluate the Safety, Tolerability and Efficacy of Single and Repeated Doses of AUP1602-C as Topical Treatment of Diabetic Foot Ulcers
Brief Title: Treatment of Diabetic Foot Ulcers With AUP1602-C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aurealis Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP-W-CLI-2018-8; 2018-003415-22 (EudraCT Number)
Record Dates: First submitted 2020-02-14; First posted 2020-02-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Analyses for phase 1 part will be done by cohort and analyses for phase 2A part will be done by treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUP1602-C (Experimental): AUP1602-C will be administered topically once or repeatedly three times per week during the treatment period.
  Interventions: Biological: AUP1602-C

INTERVENTIONS:
Biological: AUP1602-C — AUP1602-C is topically applied on chronic wounds and covered by wound dressing.

SUMMARY:
This is a two-part phase 1/2A study performed in diabetic foot ulcer (DFU) patients with chronic non-healing wounds to investigate the safety and efficacy of AUP1602-C.

DETAILED DESCRIPTION:
Study AP-W-CLI-2018-8 is the first clinical study of AUP1602-C in humans. It is a Phase 1/2A clinical study to evaluate the safety, tolerability and efficacy of a single and repeated doses of AUP-16 as topical treatment of DFU. The Phase 1 part will be a multicenter, open-label, non-randomized, uncontrolled dose-finding study with sequential dose escalations performed in dose cohorts comparing three doses of AUP-16 administered three times per week (low, medium, and high dose cohorts). This part will consist of four sequentially recruited cohorts. It is expected that a minimum of 15 patients may be required to determine the RP2D in phase 1 part.

The Phase 2A part, an extension of the Phase 1, will be a multi-center, open-label, randomized, placebo-controlled study of the recommended AUP1602-C dose and administration schedule from Phase 1 to confirm safety and to assess efficacy of the selected recommended phase 2 dose and schedule in DFU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 80 years
2. Patients with DM of type 1 or 2 having a glycosylated haemoglobin (HbA1c) of ≤11% and a serum creatinine level of ≤1.5 times the upper limit of normal (ULN)
3. Patients with at least one ulcer that fulfills all of the following criteria at screening and at baseline (prior to treatment start)

   * Present for ≥1 month
   * Located either in the plantar or on the dorsum of foot, or in the distal part of the leg, around the malleolar areato be accessible for administration of AUP1602-C/placebo and to be completely covered by the primary and secondary dressings
   * Partial- or full-thickness, not involving bone or joints, i.e. University of Texas classification Grade 1A, 1C, 2A or 2C.
   * No clinical signs of active infection or osteomyelitis
   * Size of the target ulcer for DFU must be between 1-9 cm2 after debridement
   * Chronic target ulcer, defined as <30% reduction in size in response to SoC during the 2-week screening period
   * Target ulcer appropriately debrided (<10% black and at least 50% of red/pink on a colorimetric scale)
   * Ulcer and periwound tissue suitable to using film dressings (i.e. no contraindications [e.g.: excessive exudation, maceration] and sufficient periwound space to hold the dressing)
4. Patients with more than one ulcer will be included if ulcers are separated by a minimum of 5 cm healthy tissue but only one target ulcer will be selected for the investigational treatment (based on investigator decision)
5. Patients with an ankle brachial index (ABI) ≥0.7 on the foot with the target ulcer
6. Patients with an assessment of the baseline level of neuropathy of the foot using Semmes-Weinstein monofilaments
7. Patients must adhere to wear therapeutic shoes or off-loading footwear if indicated
8. A female patient of childbearing potential must have a negative serum pregnancy test at the time of Screening
9. Patients must use a highly effective contraceptive measure (methods that can achieve a failure rate of less than 1% per year when used consistently and correctly), like hormonal contraception (oral pills, implantable device, or skin patch), intrauterine device, bilateral tubal occlusion, or double barrier throughout the study
10. Patients who understand and are willing to comply with study procedures and give written informed consent prior to enrolment in the study or initiation of study procedures

Exclusion Criteria:

1. Current or previous (within 2 weeks prior to start of screening/run-in period) treatment with another investigational drug and/or medical device or participation in another clinical study
2. Current or previous (within 30 days prior to start of screening/run-in period) treatment with a biologic agent, growth factors or skin equivalents (e.g. Regranex®, Apligraf®, or Dermagraft®)
3. Current or previous (within 2 weeks prior to first study drug dosing) treatment with active wound care agents (e.g. local and systemic antibiotics or silver dressings)
4. Current or previous (within 2 weeks prior to first study drug dosing) use of corticosteroids and immunosuppressants
5. Known hypersensitivity to any of the investigational drug or vehicle components
6. Ulcer of University of Texas Grade ≥2, with deep abscess, or gangrene
7. Target ulcer with known or suspected active infection which requires antimicrobials. Any antibiotic therapy must be completed or discontinued within 2 weeks prior to first study drug dosing
8. Target ulcer positive for MRSA
9. Target ulcer other than chronic non-healing DFU (e.g. pressure ulcers, burn wounds)
10. Prior radiation therapy (within 6 weeks prior to first study drug dosing) of any part of the foot/leg bearing the target ulcer under study
11. Sickle-cell anemia, Reynaud's, or other peripheral vascular disease including venous leg ulcers
12. Infective endocarditis or increased risk for infective endocarditis, which includes, but is not limited to, prosthetic cardiac valve or prosthetic material used for cardiac valve repair, previous infective endocarditis, congenital heart disease, and cardiac transplantation recipients who develop cardiac valvulopathy, history of rheumatic fever or rheumatic heart disease diagnosed by echocardiogram, or history (within 10 years prior to enrollment) of IV drug abuse
13. Active Charcot deformity of the study foot (i.e. foot is erythematous, warm, edematous, and is actively remodeling)
14. Patients with other reasons for wound healing disturbances: e.g. bleeding disorders, vitamin K deficiency, hypocalcemia, major immune deficiencies
15. Active malignant disease of any kind except for basal cell carcinoma (of the skin) not co-located with the target ulcer. A patient, who has had a malignant disease in the past, was treated and is currently disease-free and not on active treatment with an immune-suppressive therapy at least for 3 months, may be considered for study entry
16. Pregnant or lactating woman
17. Haemoglobin of less than 8.5 g/dL
18. Transaminase levels greater than 3 times ULN
19. Patients receiving haemodialysis or chronic ambulatory peritoneal dialysis (CAPD) therapy
20. Positive for hepatitis B or C virus (HBV, HCV), or human immunodeficiency virus (HIV); serology test results not older than 3 months are accepted
21. Planned surgery during the study period
22. Known abuse of alcohol, drugs, or medical products. Tobacco use will be allowed
23. Previous participation in this clinical study
24. Any diagnosed unstable condition that could interfere with compliance, such as psychiatric disorder
25. Myocardial infarction diagnosed within last 3 months prior to start of screening/run-in period
26. Confirmed or suspected COVID-19 infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and potential dose-limiting toxicities (DLTs) | 4 weeks
  Incidence of adverse events (AEs) and potential dose-limiting toxicities (DLTs) for safety, low, medium, and high dose cohorts of single and repeatedly administered AUP1602-C
Incidence of Treatment-Emergent Adverse Events | 6 months
  • Incidence of AEs
Incidence of Wound Closure | 6 months
  * Percentage (%) of patients with a target ulcer achieving complete wound closure
  * Percentage (%) of wound size reduction (wound area measurements in cm^2)

SECONDARY OUTCOMES:
Incidence of Wound Closure | 6 months
  * Percentage (%) of wound area (cm^2) reduction
  * Percentage (%) of wound depth (mm) reduction
  * Percentage (%) of wound volume (mm^3) reduction
  Measurements will be aggregated: Wound are and depth will be used to calculate wound volume.
Incidence of ulcer recurrence | 6 months
  Percentage (%) of patients with ulcer recurrence
Incidence of Wound Infections | 6 months
  Proportion of patients with local wound infections related to the target ulcer
Incidence of surgical procedures | 6 months
  * Number of patients with local surgical procedures
  * Incidence of amputations (minor or major) related to the target ulcer
Changes in Quality of Life according to EQ-5D-5L | 6 months
  Change from baseline in health-related quality is assessed according to EuroQoL-5 Dimensions (EQ-5D-5L) patient quesionnaire. Five single-item dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. Result of the questionnaire is scored from 0 (worst health imaginable) to 100 (best health imaginable).
Changes in Quality of Life according to DLQI | 6 months
  Change from baseline in health-related quality is assessed according to Dermatology Life Quality Index (DLQI). It consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score will be calculated as the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Changes in pain assessment according to VAS | 6 months
  Change from baseline in patient's pain intensity according to a numerical Visual Analog Scale (VAS) ranging from 0 = no pain to 10= worst imaginable pain.
Incidence of Adverse Events | 6 months
  * Incidence of abnormal vital signs
  * Incidence of abnormal ECG data
  * Incidence of abnormal echocardiogram data
  * Incidence of abnormal ophthalmoscopy data
  * Incidence of abnormal physical examination findings
  * Incidence of abnormal laboratory data
Incidence of bacteria distribution | 6 months
  Assessment of biodistribution and shedding (yes / no)

CONTACTS AND LOCATIONS:
Locations (2):
- Medizinische Hochschule Hannover (MHH) CRC Core Facility, Hanover, Germany
- Mikomed, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schindler C, Mikosinski J, Mikosinski P, Karkkainen HR, Sanio M, Kurkipuro J, Mierau I, Smith W, Vartiainen A, Decory L, Weber D, Wirth T, Yrjanheikki J, Schellong S, Samaranayake H. Multi-target gene therapy AUP1602-C to improve healing and quality of life for diabetic foot ulcer patients: a phase I, open-label, dose-finding study. Ther Adv Endocrinol Metab. 2024 Nov 4;15:20420188241294134. doi: 10.1177/20420188241294134. eCollection 2024. PMID 39838970